CLINICAL TRIAL: NCT03766620
Title: A Prospective, Observational Study, of a High Calorie, High Protein Tube Feeding With Slow Release Carbohydrates and Monounsaturated Fatty Acids (MUFA), in a Malnourished Population With Diabetes
Brief Title: A Tube Feeding Study in Malnourished Population With Diabetes
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA14
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Malnutrition; Diabetes
MeSH Terms: conditions — Malnutrition; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tube Fed Participants: Individuals with diabetes and malnutrition receiving tube feed as sole source nutrition.

SUMMARY:
This is a prospective, non-interventional, observational study. Malnourished subjects with diabetes, who are receiving a high calorie, high protein tube feeding with slow release carbohydrates and MUFA by their health care professional (HCP) per standard of care will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated an informed consent form, approved by an Independent Ethics Committee, prior to any participation in the study
* Considered malnourished, or at risk for malnutrition
* Diagnosed with diabetes mellitus type 1 or 2 and treated with oral hypoglycemic medications and/or exogenous insulin
* Conforms to the requirements set forth on the study product label
* Under the care of a health care professional for malnutrition and has recently been prescribed tube feeding as a sole-source of nutrition by their health care professional
* Free living, residing in a nursing home or admitted to the hospital and has anticipated length of hospital stay > 3 days and < 12 days

Exclusion Criteria:

* Severe dementia or delirium, eating disorder, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Cannot safely consume the study product, or known to be allergic or intolerant to any ingredient found in the study product
* Renal or liver failure
* Participates in another study that has not been approved as a concomitant study by AN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects, men and women who meet all enrollment criteria, will be enrolled from study centers in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Body Weight Change | Baseline to Study Exit Week 12
  Measured in Kg

SECONDARY OUTCOMES:
Malnutrition Universal Screening Tool (MUST) | Baseline to Study Exit Week 12
  HCP completed screening tool
Subjective Global Assessment (SGA) | Baseline to Study Exit Week 12
  HCP completed nutrition assessment
Quality of life (EuroQol EQ-5D-5L) | Baseline to Study Exit Week 12
  Subject rated health state of 5 dimensions. Each dimension has 5-levels scaled in negative direction resulting in an overall 5-digit number describing the health state; EQ VAS Score 0-100 points scaled in positive direction
Glucose control | Baseline to Study Exit Week 12
  HbA1c levels
Body Mass Index | Baseline to Study Exit Week 12
  BMI calculated Weight (kg)/Height (m)2
Product Compliance | Baseline to Study Exit Week 12
  Product consumption diary
Albumin Levels | Baseline to Study Exit Week 12
  Nutrition status parameter collected per standard of care

OTHER OUTCOMES:
Functionality | Baseline to Study Exit Week 12
  Barthel Index of Activities of Daily Living; Subject completed assessment of 10 functions; Sum of scores range from 0-20 scaled in positive direction
Physician Product Satisfaction | Baseline to Study Exit Week 12
  Physician Completed Questionnaire; 3 to 5 category responses scaled in negative direction

CONTACTS AND LOCATIONS:
Overall Officials: Maria Camprubi Robles, PhD, Study Chair — Abbott; Angela M Palmero, MD, Study Chair — Hospital San Pedro de La Rioja
Locations (8):
- Spain (8):
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Costa del Sol 3095, Marbella, Málaga
  - Hospital Costa del Sol 3178, Marbella, Málaga
  - Hospital Universitario La Paz, Madrid
  - Hospital Gomez-Ulla, Madrid
  - Centro Médico San juan de la Cruz, Málaga
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided